CLINICAL TRIAL: NCT02382991
Title: Randomized, Cross-over Study Comparing the Efficacy of the 3C60 Knee Against Non-microprocessor Controlled Knees on the Risk of Falling and Locomotor Skills of Moderately Active Persons With Leg Amputation Above Knee or Knee Disarticulation
Brief Title: Assessment of Disability Compensation With the C-LEG COMPACT 2 Knee (Ref. 3C60 et 3C60=ST)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Bock France SNC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20PT002-FR-01-0614; 2014-A00754-43 (Registry Identifier: RCB (ANSM))
Record Dates: First submitted 2015-02-25; First posted 2015-03-09 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-09

CONDITIONS: Amputation of Hip and Thigh, Level Unspecified
Keywords: Moderately active amputees; C-leg Compact; Knee prosthesis; Kenevo; Microprocessor controlled knee; Amputation; 3C60; Timed Get Up and Go (TGUG); Locomotors Capacities Index (LCI); QUEST; Short Form survey (SF-36)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NMPK-3C60 (Other): D0 + 30 days: evaluation with the non-microprocessor knee. D1 + 90 days: evaluation with the 3C60 knee.
  Interventions: Device: 3C60-NMPK
- 3C60-NMPK (Other): D0 + 90 days: evaluation with the 3C60 knee. A period of 10 days of "wash out". D1 + 30 days: evaluation with the non-microprocessor knee.
  Interventions: Device: NMPK-3C60

INTERVENTIONS:
Device: 3C60-NMPK — 3 months with 3C60 - 10 days wash out - 1 month with NMPK
  Other Names: Mechanical knee joint
  Arms: NMPK-3C60
Device: NMPK-3C60 — 1 month with NMPK - 3 months with 3C60
  Other Names: C-LEG COMPACT 2; KENEVO
  Arms: 3C60-NMPK

SUMMARY:
Moderately active amputees may have lost their limb due to diabetes, vascular conditions, trauma, tumour or congenital causes. These amputees currently cannot benefit from having a computerised knee because of the performance criteria associated with being given one. However, these amputees have a very high risk of falling because they use a non microprocessor controlled knee joint (NMPK) and because their physical ability, associated disability and persistent contralateral leg weakness do not allow them to compensate for a balance deficit. These amputees restrict how much they move around and their participation because of their instability and elevated risk of falling.

The objective of the study is to evaluate the effect of the 3C60 knee, a microprocessor-controlled knee joint for external leg prosthesis, on the reduction in the risk of falling after three months in moderately active persons with leg amputation above knee or knee disarticulation.

DETAILED DESCRIPTION:
The patient will be evaluated after one month of using his/her usual non micropressor controlled knee joint (NMPK). After fitting of the 3C60, the patient will undergo at least five rehabilitation sessions, adapted to his/her individual needs, so that he/she knows how to use the device and is ready to go along with the planned testing.

After the trial with the 3C60 knee, the patient will again be fitted with his/her non microprocessor controlled knee joint (NMPK) and will be required to undergo one rehabilitation session to regain his/her walking abilities.

ELIGIBILITY:
Inclusion Criteria:

* Person with leg amputation above knee or knee disarticulation with stabilized residual limb
* Person who are currently fitted with a prosthesis using a non-microprocessor controlled prosthetic knee
* Person with a high risk of falling, which is defined as a TGUG test score of more than 19 seconds
* Person who moves around within buildings other than one's residence, such as moving around other people's homes, other private buildings, community and private or public buildings and enclosed areas, moving throughout all parts of buildings and enclosed areas, between floors, inside, outside and around buildings, both public and private
* Person who moves around outside the home and other buildings, such as walking and moving around close to or far from one's home and other buildings, without the use of transportation, public or private, such as walking for short or long distances around a town or village, walking or moving down streets in the neighbourhood, town, village or city; moving between cities and further distances, without using transportation
* Person with a daily walking distance greater than 300 m

Exclusion Criteria:

* Persons using underarm crutches or walkers
* Persons under 18 years of age
* Persons who weigh more than 125 kg
* Pregnant women
* Persons in an emergency situation
* Persons who cannot personally provide their consent
* Persons who are not available to follow the entire study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Chiesa, Physician, Principal Investigator — Institut Robert Merle d'Aubigné - 2 rue du Parc 94460 Valenton - France
Locations (15):
- Sonderkrankenanstalt Zicksee, Sankt Andrä am Zicksee, Austria
- France (13):
  - CRMPR "Les Herbiers", Bois-Guillaume
  - Hôpital d'instruction des Armées Percy, Clamart
  - Centre Hospitalier de Cornouaille Concarneau, Concarneau
  - Centre de réadaptation de Coubert, Coubert
  - CHU de Grenoble Hôpital Sud, Échirolles
  - Clinique Chantecler, Marseille
  - Institut Régional de Médecine Physique et de Réadaptation, Nancy
  - Institut National des Invalides, Paris
  - Hôpital Léopold Belan, Paris
  - Pôle Saint-Hélier, Rennes
  - Hôpital privé de l'Est Lyonnais, Saint-Priest
  - Centre l'Adapt Thionis, Thionville
  - Institut Robert Merle d'Aubigné, Valenton
- Universitätsmedizin Göttingen, Göttingen, Germany

REFERENCES:
- [Background] Schoppen T, Boonstra A, Groothoff JW, de Vries J, Goeken LN, Eisma WH. The Timed "up and go" test: reliability and validity in persons with unilateral lower limb amputation. Arch Phys Med Rehabil. 1999 Jul;80(7):825-8. doi: 10.1016/s0003-9993(99)90234-4. PMID 10414769
- [Background] Dite W, Connor HJ, Curtis HC. Clinical identification of multiple fall risk early after unilateral transtibial amputation. Arch Phys Med Rehabil. 2007 Jan;88(1):109-14. doi: 10.1016/j.apmr.2006.10.015. PMID 17207685
- [Background] Franchignoni F, Orlandini D, Ferriero G, Moscato TA. Reliability, validity, and responsiveness of the locomotor capabilities index in adults with lower-limb amputation undergoing prosthetic training. Arch Phys Med Rehabil. 2004 May;85(5):743-8. doi: 10.1016/j.apmr.2003.06.010. PMID 15129398
- [Background] Gauthier-Gagnon C, Grise MC, Potvin D. Enabling factors related to prosthetic use by people with transtibial and transfemoral amputation. Arch Phys Med Rehabil. 1999 Jun;80(6):706-13. doi: 10.1016/s0003-9993(99)90177-6. PMID 10378500
- [Background] Burnfield JM, Eberly VJ, Gronely JK, Perry J, Yule WJ, Mulroy SJ. Impact of stance phase microprocessor-controlled knee prosthesis on ramp negotiation and community walking function in K2 level transfemoral amputees. Prosthet Orthot Int. 2012 Mar;36(1):95-104. doi: 10.1177/0309364611431611. Epub 2012 Jan 5. PMID 22223685
- [Background] Gauthier-Gagnon, C, grisé, MCL, Lepage Y. The Locomotor Capabilities Index : Content validity. J rehabil OutcomesMeas 2(4) : 40-46, 1998.
- [Background] Gauthier-Gagnon, C, Grisé, MCL, Potvin, L. Predisposing factors related to prosthetic use by people with a transtibial and transfemoral amputation. J Prosthet Orthot 10: 99-109, 1998
- [Background] Gauthier-Gagnon C, Grise MC. Prosthetic profile of the amputee questionnaire: validity and reliability. Arch Phys Med Rehabil. 1994 Dec;75(12):1309-14. PMID 7993169
- [Background] Grise MC, Gauthier-Gagnon C, Martineau GG. Prosthetic profile of people with lower extremity amputation: conception and design of a follow-up questionnaire. Arch Phys Med Rehabil. 1993 Aug;74(8):862-70. doi: 10.1016/0003-9993(93)90014-2. PMID 8347072
- [Background] Demers L, Weiss-Lambrou R, Ska B. Development of the Quebec User Evaluation of Satisfaction with assistive Technology (QUEST). Assist Technol. 1996;8(1):3-13. doi: 10.1080/10400435.1996.10132268. PMID 10159726
- [Background] Leplege A, Mesbah M, Marquis P. [Preliminary analysis of the psychometric properties of the French version of an international questionnaire measuring the quality of life: the MOS SF-36 (version 1.1)]. Rev Epidemiol Sante Publique. 1995;43(4):371-9. French. PMID 7667543
- [Background] Leplège, A. (2001). Introduction, enjeux, définitions. In J. Coste et A. Leplège (Eds.), Mesure de la santé perceptuelle et de la qualité de vie : méthodes et applications (pp 15-36). Paris : Editions Estem
- [Background] Ware JE, Snow KK, Kosinski M, Gandek B (1993). Health survey : manual and interpretation guide. Boston, Massachussets : The Health Institute, New England Medical Center, 1993
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Loiret I, Paysant J, Martinet N, Andre JM. [Evaluation of amputees]. Ann Readapt Med Phys. 2005 Jul;48(6):307-16. doi: 10.1016/j.annrmp.2005.03.009. Epub 2005 Apr 15. French. PMID 15932782

RESULTS

PARTICIPANT FLOW:
Groups:
- NMPK (30 Days), 3C60 (90 Days): D0 + 30 days: evaluation with the non-microprocessor knee. D1 + 90 days: evaluation with the 3C60 knee.
  3C60-NMPK: 3 months with 3C60 - 10 days wash out - 1 month with NMPK
- 3C60 (90 Days), Washout (10 Days), NMPK (30 Days): D0 + 90 days: evaluation with the 3C60 knee. A period of 10 days of "wash out". D1 + 30 days: evaluation with the non-microprocessor knee.
  NMPK-3C60: 1 month with NMPK - 3 months with 3C60
Period: Overall Study
Arm/Group | NMPK (30 Days), 3C60 (90 Days) | 3C60 (90 Days), Washout (10 Days), NMPK (30 Days)
Started | 17 | 18
Completed | 15 | 15
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group NMPK Then 3C60: This arm group includes 17 participants who were first fitted with Non MicroProcessor-controlled Knee (30 days) then with 3C60 knee (90 days).
- Group 3C60 Then NMPK: This arm group includes 18 participants who were first fitted with 3C60 knee (90 days) then had a washout period (10 days) then where fitted with Non MicroProcessor-controlled Kne (30 days).
- Total: Total of all reporting groups
Arm/Group | Group NMPK Then 3C60 | Group 3C60 Then NMPK | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] — The Age of the participants was recorded at baseline. This was meant for describing the population. No value was considered better or worse outcome.
  years | 66.94 (9.6) | 63.28 (10.5) | 65.06 (10.1)
Sex/Gender, Customized [Number; unit: Percentage of participants] — The sexe of the participants was recorded at baseline. This was meant for describing the population. No value was considered better or worse outcome.
  Percentage of participants
    Male | 76.5 | 77.8 | 77.1
    Female | 23.5 | 22.2 | 22.9
Amputation cause [Number; unit: Percentage of participants] — Amputation cause was recorded at baseline. This was meant for describing the population. No amputation cause was considered better or worse outcome.
  Percentage of participants
    Vascular | 35.3 | 55.6 | 45.7
    Vascular diabetic | 11.8 | 11.1 | 11.4
    Traumatic | 23.5 | 22.2 | 22.9
    Tumour | 11.8 | 11.1 | 11.4
    Infectious | 17.6 | 0 | 8.6
Amputation level [Number; unit: Percentage of participants] — Amputation level was recorded at baseline. This was meant for describing the population. No amputation level was considered better or worse outcome.
  Percentage of participants
    Transfemoral | 94.1 | 94.4 | 94.3
    Knee disarticulation | 5.9 | 5.6 | 5.7
Weight [Mean (Standard Deviation); unit: Kg] — Participants' weight was recorded at Baseline. This was meant for describing the population. No value was considered better or worse outcome.
  Kg | 76.1 (16.6) | 76.2 (16.2) | 76.1 (16.1)
Height [Mean (Standard Deviation); unit: cm] — Height of the participants was recorded at baseline. This was meant for describing the population. No value was considered better or worse outcome.
  cm | 170.3 (10.2) | 172.3 (7.7) | 171.3 (8.6)
Time since amputation [Mean (Standard Deviation); unit: months] — Time since amputation was recorded at baseline. This was meant for describing the population. No value was considered better or worse outcome.
  months | 51.3 (62.1) | 70.8 (105.1) | 61.4 (85.5)
International Classification of Function (ICF) [Number; unit: Percentage of participants] — International Classification of Functioning was recorded at baseline. This was meant for describing the population. No mobility grade was considered better or worse outcome.
  d4602: Moving around outside the home and other buildings d4601: Moving around within buildings other than home
  Percentage of participants
    d4602 | 94.1 | 88.9 | 91.4
    d4601 | 5.9 | 11.1 | 8.6
Additional disabilities [Number; unit: Percentage of participants] — Additional disabilities were recorded at baseline. This was meant for describing the population. No data was considered better or worse outcome.
  Percentage of participants
    Trans-tibial amputation of the controlateral lower | 2.9 | 11.1 | 8.6
    forefoot amputation on the controlateral side | 2.9 | 0 | 2.9
    Handicap of the upper limbs | 0 | 11.1 | 5.7
    Traumatism of the controlateral lower limb | 2.9 | 0 | 2.9
    Hemiplegia after a stroke affecting balance | 0 | 5.6 | 2.9
Geographical area [Number; unit: Percentage of participants] — Geographical area was recorded at baseline. This was meant for describing the population. No data was considered better or worse outcome.
  Percentage of participants
    Urban | 70.6 | 66.7 | 68.6
    Rural | 29.4 | 33.3 | 31.4
work status [Number; unit: Percentage of participants] — Work status was recorded at baseline. This was meant for describing the population. No data was considered better or worse outcome.
  Percentage of participants
    With a professional activity | 0 | 11.1 | 5.7
    Without activity | 23.5 | 22.2 | 22.9
    Retired | 76.5 | 66.7 | 71.4
previous prosthesis [Number; unit: Percentage of participants] — Type of knee on the previous prosthesis was recorded at baseline. This was meant for describing the population. No data was considered better or worse outcome.
  Percentage of participants
    Locked knee | 29.4 | 38.9 | 34.3
    Brake knee | 17.6 | 16.7 | 17.1
    Pneumatic knee | 17.6 | 5.6 | 11.4
    Hydraulic knee | 29.4 | 33.3 | 31.4
    Free knee | 5.9 | 5.6 | 5.7
socket type [Number; unit: Percentage of participants] — Socket type was recorded at baseline. This was meant for describing the population. No data was considered better or worse outcome.
  Percentage of participants
    Quadrangular | 0 | 5.6 | 2.9
    With ischial containment | 88.2 | 88.9 | 88.6
    For knee disarticulation | 5.9 | 5.6 | 5.7
prosthetic foot with mechanical knee [Number; unit: Percentage of participants] — Prosthetic foot on the previous prosthesis was recorded at baseline. This was meant for describing the population. No foot type was considered better or worse outcome.
  Percentage of participants
    Dynamic with carbon | 41.2 | 50.0 | 45.7
    Dynamic without carbon | 29.4 | 22.2 | 25.7
    Articulated | 17.6 | 16.7 | 17.1
    Solid Ankle Cushion Heel (SACH) | 11.8 | 11.1 | 11.4

OUTCOME MEASURES:

1. Primary Outcome: Timed Get Up and Go (TGUG)
Description: This test consists of recording the amount of time needed for a person to stand up from a chair, walk 3 metres, make a half-turn and sit down again. The TGUG test score reflects a person's balance and as a consequence, the risk of falling.
Time Frame: Measurement will be performed at 3 months with 3C60 and at 1 month with NMPK
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Overall
Number analyzed (Participants) | 30
seconds
  NMPK | 24.8 (8.3)
  3C60 | 21.6 (9.0)

2. Secondary Outcome: Locomotor Capabilities Index (LCI-5)
Description: The Locomotor Capabilities Index (LCI-5) is a 14 item self-assessment questionnaire filled in by the patient that explores walking and ambulation. The LCI-5 is derived from the Prosthesis Profile of the Amputee Questionnaire (PPA). LCI-5 is sensitive to the use of walking aids or to the need of a third party. Ceiling effect is not expected with moderately active amputees. The global LCI-5 score is the addition of the 14 scores, noted between 0 and 4. The global score varies between 0 and 56, the highest being for persons with high locomotors capabilities. LCI-5 has two sub-scores: the basic score corresponds to 7 questions related to basic activities and the advanced score corresponds to 7 questions related to more advanced activities. The basic and advanced scores both range from 0-28. Higher scores correspond with a better outcome.
Time Frame: Measurement will be performed at 3 months with 3C60 and at 1 month with NMPK
Measure: Mean (Standard Deviation); unit: Score between 0 and 56
Arm/Group | Overall
Number analyzed (Participants) | 30
Score between 0 and 56
  NMPK - Global score | 38.6 (9.5)
  3C60 - Global score | 41.7 (7.3)
  NMPK - Basic score | 20.1 (4.8)
  3C60 - Basic score | 21.9 (3.8)
  NMPK - Advances score | 18.5 (5.5)
  3C60 - Advanced score | 19.8 (5.0)

3. Secondary Outcome: Use of Walking Aids
Description: The type of walking aids used with each device will be recorded.
Time Frame: Measurement will be performed at 3 months with 3C60 and at 1 month with NMPK
Population: No significant difference in the repartition of walking aids was - a priori- expected between both devices: NMPK and 3C60.
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 30
participants
  NMPK - none | 7
  3C60 - none | 7
  NMPK - 1 cane | 7
  3C60 - 1 cane | 7
  NMPK - 1 crutch | 3
  3C60 - 1 crutch | 5
  NMPK - 2 canes | 3
  3C60 - 2 canes | 3
  NMPK - 2 crutches | 9
  3C60 - 2 crutches | 8
  NMPK - Walking frame | 1
  3C60 - walking frame | 0

4. Secondary Outcome: QUEST 2.0 Satisfaction Questionnaire (QUEST 2.0-G: German Version / ESAT: French Version)
Description: It is a self-evaluation questionnaire of the user's satisfaction, translated in French (ESAT) and in German (QUEST 2.0-G Section 17.5). The QUEST 2.0 questionnaire contains 8 items that evaluate the device's technology and 4 items that evaluate services surrounding the device. It allows patients to express themselves on the criteria that are most important to them. Each item has a score that varies between 0 (not satisfied at all) and 5 (very satisfied). The global score is the average obtained onto the 12 items. Two sub-scores related to the technology and services can also be calculated. They correspond to the average of the 8 first items and to the 4 last items respectively. All scores ranks between 0 and 5, 5 being the highest level of satisfaction.
Time Frame: Measurement will be performed at 3 months with 3C60 and at 1 month with NMPK
Measure: Mean (Standard Deviation); unit: Score from 0 to 5
Arm/Group | Overall
Number analyzed (Participants) | 30
Score from 0 to 5
  NMPK - Global score | 3.7 (0.8)
  3C60 - Global score | 4.4 (1.0)
  NMPK - Services | 4.1 (0.7)
  3C60 - Services | 4.5 (1.1)
  NMPK - Technology | 3.7 (0.8)
  3C60 - Technology | 4.3 (0.8)

5. Secondary Outcome: SF-36v2™ Health Survey
Description: 36-Item Short Form Health Survey (SF-36v2TM) explores 8 dimensions of quality of life through 36 questions: PF= Physical Functioning (10 items), RP= Role Physical (4 items), BP = Bodily Pain (2 items), SF= Social Functioning (2 items), MH= Mental Health (5 items), RE= Role emotional (3 items), VT= Vitality (4 items), GH= General Health (5 items). All of the eight health domain scales contributes with different levels to score two component summary measures: PCS= Physical Component Summary and MCS= Mental Component Summary. All scores are calculated online through scoring software. Domain scales and component summary are ranging from 0 to 100. A high score is considered to be a better outcome, as indicating little or no problem.
Time Frame: Measurement will be performed at 3 months with 3C60 and at 1 month with NMPK
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Overall
Number analyzed (Participants) | 30
scores on a scale
  NMPK - Physical Component Score | 43.1 (6.7)
  3C60 - Physical Component Score | 45.0 (8.4)
  NMPK - Mental Component Score | 56.6 (9.7)
  3C60 - Mental Ccomponent Score | 56.0 (7.3)

6. Secondary Outcome: Number of Falls
Time Frame: Measurement will be performed at 1 month with both devices
Measure: Number; unit: falls
Arm/Group | Overall
Number analyzed (Participants) | 30
falls
  NMPK - number of falls occured | 6
  3C60 - number of falls occured | 1
  NMPK - number related to the knee | 4
  3C60 - number related to the knee | 0

ADVERSE EVENTS:
Groups:
- NMPK: Participants with non microprocessor-controlled knee joint
- 3C60: Participants with 3C60 knee joint
Arm/Group | NMPK | 3C60
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/35
Other Adverse Events (participants affected / at risk) | 2/35 | 10/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NMPK (N=35) | 3C60 (N=35)
Hospitalization due to other reason than amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NMPK (N=35) | 3C60 (N=35)
Non serious adverse events related to the knee (Social circumstances) | 2 (4) | 2 (2)
Non serious adverse events maybe related to the knee (Social circumstances) | 0 (0) | 3 (3)
Non serious adverse events not related to the knee (Social circumstances) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No